CLINICAL TRIAL: NCT00223717
Title: The Pathophysiology and Treatment of Supine Hypertension in Patients With Autonomic Failure
Brief Title: Treatment of Supine Hypertension in Autonomic Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 010189
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
Keywords: Supine Hypertension; Hypertension; Treatment; Autonomic failure; Pure autonomic failure; Multiple System Atrophy; Shy-Drager Syndrome
MeSH Terms: conditions — Hypertension; Pure Autonomic Failure; Multiple System Atrophy; Shy-Drager Syndrome | interventions — Clonidine; Nitroglycerin; Dipyridamole; Aspirin; Aspirin, Dipyridamole Drug Combination; Deamino Arginine Vasopressin; Sildenafil Citrate; Nifedipine; Hydralazine; Hydrochlorothiazide; Bosentan; Diltiazem; Eplerenone; Guanfacine; Arginine; Captopril; Carbidopa; Losartan; Metoprolol; Nebivolol; Prazosin; Tamsulosin; aliskiren

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Active drug or intervention (Experimental): Clonidine, Nitroglycerin transdermal, Dipyridamole/ Aspirin (Aggrenox), Desmopressin (DDAVP), Sildenafil, Nifedipine, Hydralazine, Hydrochlorothiazide, Bosentan, Diltiazem, Eplerenone, guanfacine, L-arginine, captopril, carbidopa, losartan, metoprolol tartrate, nebivolol hydrochloride, prazosin hydrochloride, tamsulosin hydrochloride, Head-up tilt, aliskiren, local heat stress
  Interventions: Drug: Clonidine; Drug: Nitroglycerin transdermal; Drug: Dipyridamole/ Aspirin (Aggrenox); Drug: Desmopressin (DDAVP); Drug: Sildenafil; Drug: Nifedipine; Drug: Hydralazine; Drug: Hydrochlorothiazide; Drug: Bosentan; Drug: Diltiazem; Drug: Eplerenone; Drug: guanfacine; Dietary Supplement: L-arginine; Drug: captopril; Drug: carbidopa; Drug: losartan; Drug: metoprolol tartrate; Drug: nebivolol hydrochloride; Drug: prazosin hydrochloride; Drug: tamsulosin hydrochloride; Other: Head-up tilt.; Drug: aliskiren; Other: Local heat stress
- 2: Placebo (Placebo Comparator): placebo pill or patch
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — 0.1-0.2mg po. Single dose.
  Other Names: Catapres
  Arms: 1: Active drug or intervention
Drug: Nitroglycerin transdermal — 0.05-0.2 mg patch. 1 application. Alone or in combination with DDAVP.
  Other Names: Nitro-Dur
  Arms: 1: Active drug or intervention
Drug: Dipyridamole/ Aspirin (Aggrenox) — dipyridamole 200 mg and aspirin 25 mg po. Single dose.
  Other Names: Aggrenox
  Arms: 1: Active drug or intervention
Drug: Desmopressin (DDAVP) — 0.2 - 0.6mg po. Single dose. Alone or in combination with nitroglycerin transdermal or nifedipine
  Other Names: DDAVP
  Arms: 1: Active drug or intervention
Drug: Sildenafil — 25- 100 mg po. Single dose.
  Other Names: Viagra
  Arms: 1: Active drug or intervention
Drug: Nifedipine — 10-30 mg po. Single dose.
  Other Names: Adalat
  Arms: 1: Active drug or intervention
Drug: Hydralazine — 10-50 mg po. Single dose
  Arms: 1: Active drug or intervention
Drug: Hydrochlorothiazide — 12.5-100 mg po. Single dose.
  Other Names: Microzide
  Arms: 1: Active drug or intervention
Drug: Placebo — Po or patch. Single dose.
  Arms: 2: Placebo
Drug: Bosentan — 62.5 -125 mg po. Single dose.
  Other Names: Tracleer
  Arms: 1: Active drug or intervention
Drug: Diltiazem — 30-60 mg po. Single dose.
  Other Names: Cardizem
  Arms: 1: Active drug or intervention
Drug: Eplerenone — 50-100 mg po. Single dose.
  Other Names: Inspra
  Arms: 1: Active drug or intervention
Drug: guanfacine — 1-3 mg po. Single dose.
  Other Names: Tenex
  Arms: 1: Active drug or intervention
Dietary Supplement: L-arginine — 6-17 g po. Single dose
  Arms: 1: Active drug or intervention
Drug: captopril — 25-50 mg PO. Single dose.
  Other Names: capoten
  Arms: 1: Active drug or intervention
Drug: carbidopa — 25-200 mg PO. Single dose.
  Other Names: Lodosyn
  Arms: 1: Active drug or intervention
Drug: losartan — 25-200 mg PO. Single dose.
  Other Names: cozaar
  Arms: 1: Active drug or intervention
Drug: metoprolol tartrate — 25-100 mg PO. Single dose.
  Other Names: lopressor
  Arms: 1: Active drug or intervention
Drug: nebivolol hydrochloride — 2.5-40 mg PO. Single dose.
  Other Names: Bystolic
  Arms: 1: Active drug or intervention
Drug: prazosin hydrochloride — 0.5-1 mg PO. Single dose.
  Other Names: Minipress
  Arms: 1: Active drug or intervention
Drug: tamsulosin hydrochloride — 0.4-0.8 mg PO. Single dose.
  Other Names: Flomax
  Arms: 1: Active drug or intervention
Other: Head-up tilt. — Head of the bed elevated 10 degrees (7 inch) or whole bed tilted head-up 5 degrees in reverse trendelenburg (head of the bed elevated 7 inches)
  Other Names: HUT
  Arms: 1: Active drug or intervention
Drug: aliskiren — aliskiren (Tekturna) 150-300mg po single dose
  Other Names: Tekturna
  Arms: 1: Active drug or intervention
Other: Local heat stress — Passive heat-stress using a commercial heating pad applied over the abdomen and part of the torso
  Other Names: heating pad
  Arms: 1: Active drug or intervention

SUMMARY:
Supine hypertension is a common problem that affects at least 50% of patients with primary autonomic failure. Supine hypertension can be severe, and complicates the treatment of orthostatic hypotension. Drugs used for the treatment of orthostatic hypotension (eg, fludrocortisone and pressor agents), worsen supine hypertension. High blood pressure may also cause target organ damage in this group of patients. The pathophysiologic mechanisms causing supine hypertension in patients with autonomic failure have not been defined.

In a study, we, the investigators at Vanderbilt University, examined 64 patients with AF, 29 with pure autonomic failure (PAF) and 35 with multiple system atrophy (MSA). 66% of patients had supine systolic (systolic blood pressure [SBP] > 150 mmHg) or diastolic (diastolic blood pressure [DBP] > 90 mmHg) hypertension (average blood pressure [BP]: 179 ± 5/89 ± 3 mmHg in 21 PAF and 175 ± 5/92 ± 3 mmHg in 21 MSA patients). Plasma norepinephrine (92 ± 15 pg/mL) and plasma renin activity (0.3 ± 0.05 ng/mL per hour) were very low in a subset of patients with AF and supine hypertension. (Shannon et al., 1997).

Our group has showed that a residual sympathetic function contributes to supine hypertension in patients with severe autonomic failure and that this effect is more prominent in patients with MSA than in those with PAF (Shannon et al., 2000). MSA patients had a marked depressor response to low infusion rates of trimethaphan, a ganglionic blocker; the response in PAF patients was more variable. At 1 mg/min, trimethaphan decreased supine SBP by 67 +/- 8 and 12 +/- 6 mmHg in MSA and PAF patients, respectively (P < 0.0001). MSA patients with supine hypertension also had greater SBP response to oral yohimbine, a central alpha2 receptor blocker, than PAF patients. Plasma norepinephrine decreased in both groups, but heart rate did not change in either group. This result suggests that residual sympathetic activity drives supine hypertension in MSA; in contrast, supine hypertension in PAF.

It is hoped that from this study will emerge a complete picture of the supine hypertension of autonomic failure. Understanding the mechanism of this paradoxical hypertension in the setting of profound loss of sympathetic function will improve our approach to the treatment of hypertension in autonomic failure, and it could also contribute to our understanding of hypertension in general.

DETAILED DESCRIPTION:
1. Overnight Medication Trials:

   Patients will be studied on the GCRC while in 150 mEq/day sodium balance and on a diet free of substances which interfere with catecholamine determination. Subjects will be asked to use the bathroom to empty their bladder at 8:00 PM. They will be given a randomly chosen medication aliskiren (Tekturna) 150-300mg po, bosentan (Tracleer) 62.5 -125 mg po, captopril 25-50mg po, carbidopa 25-200mg po, clonidine 0.1-0.2mg po, desmopressin 0.2 - 0.6mg po (DDAVP), -diltiazem 30-60 mg po, dipyridamole 200 mg and aspirin 25 mg po (Aggrenox), eplerenone (Inspra) 50-100 mg po, guanfacine (Tenex) 1-3 mg po, hydralazine 10-50 mg po, hydrochlorothiazide 12.5-100 mg po, L- arginine 6-17 g po, losartan 25-100mg po, metoprolol tartrate (Lopressor) 25-100 mg po, nebivolol hydrochloride (Bystolic) 2.5-40 mg po, nitroglycerin-transdermal 0.05-0.2 mg patch, nifedipine (adalat) doses 10-30 mg, prazosin hydrochloride 0.5-1 mg po, sildenafil (Viagra) 25- 100 mg po, tamsulosin hydrochloride (Flomax) 0.4-0.8 mg po. The combination desmopressin 0.2 mg po (DDAVP) and nitroglycerin-transdermal 0.05-0.2 mg. The combinations desmopressin 0.2 mg po and nifedipine (10-30 mg). A placebo pill or skin patch will be done as a control to measure their supine blood pressure without medication intervention. They will then be asked to lie down with the head of the bed elevated 10 degrees. An automated blood pressure cuff (Dinamap) will be wrapped around an upper arm and blood pressure will be measured automatically 2 times in a row every 2 hours. At 8 AM the following morning the study ends. The subjects will then stand at the bedside as motionless as possible for 30 minutes for blood pressure and heart rate determination.

   Urine will be collected for 24 hours for determination of volume and sodium, potassium and catecholamines (for some medication trials) in 12 hour segments, from 8 a.m. to 8 p.m. and 8 p.m. to 8 a.m. to ascertain how the medications affect urine production.

   For medication trials affecting renal Na and/or water regulation (e.g. desmopressin, carbidopa), blood samples will be collected (5 mL, 1 teaspoon) at 8 PM and 8 AM for determination of a basic metabolic panel.

   Raising the head of the bed during the night is a non-pharmacologic measure that may reduce supine blood pressure, nocturnal natriuresis and improve orthostatic hypotension the following morning in autonomic failure patients with supine hypertension. However, it is not known if tilting the bed with the head up is better than raising only the head of the bed. To compare the effect of these two ways of raising the head of the bed on nighttime blood pressure and nocturnal natriuresis, some patients will undergo two additional tests. On two separate nights (either consecutive or not), patients will receive the placebo and will be assigned by simple randomization to lie down in one of two different bed positions:
   1. The head of the bed elevated 10 degrees (~ 7 inches); or
   2. The whole bed tilted head-up 5 degrees in reverse trendelenburg (head of the bed elevated ~7 inches).

   Blood pressure, orthostatic tolerance at 8 AM and urine collections will be performed as described above.
2. Blood Pressure Lowering Effect of Local Heat Stress in Supine Hypertension:

   Heat stress due to high environmental temperatures lowers blood pressure in autonomic failure patients. The mechanisms underlying this phenomenon are not fully understood but it could be associated with 2 factors: First, heart stress is more likely to increase core temperature in this patient population because heat dissipation is impaired due to inability to sweat. Second, autonomic failure patients lack the compensatory sympathetic splanchnic vasoconstriction and tachycardia that normally maintain blood pressure in response to heat stress in healthy subjects. We hypothesize, therefore, that even moderate levels of local heat stress will lower blood pressure in patients with autonomic failure and supine hypertension. We propose a pilot study to evaluate the effect of local (abdominal) heat stress on blood pressure in autonomic failure patients, something that has not been previously done, and to assess its potential use in the treatment of supine hypertension

   This pilot study is optional and will be conducted in patients already enrolled in the "Evaluation and Treatment of Autonomic Failure" and the medication trial part of this protocol. Subjects will be studied in the supine position on two study days (with and without heat stress). Each study day will last ~3 hours. Core body and skin temperature will be monitored throughout the study using an ingestible telemetry pill and dermal patches. Blood pressure and heart rate will be measured intermittently with an automated blood pressure sphygmomanometer wrapped around an upper arm. Segmental body fluid shifts will be estimated using bioelectrical Impedance and hemodynamic parameters using body impedance and the rebreathing test (Innocor). After obtaining normothermic baseline measurements, we apply passive heat-stress with a commercial heating pad that covers all the abdomen and part of the torso to provide local heating at ~44ºC continuously for 2 hr. Outcome measurements are obtained at 1 and 2 hours after passive heat-stress, or when the CBT increases ~1ºC above baseline, whichever occurs first. For the control (non-heating) study day, the heating pad will be applied on patients but we will not turn it on, and data collection will be performed at the one-hour intervals for 2 hours, to provide a time control.
3. Circadian Hemodynamic Changes in Autonomic Failure Patients with Supine Hypertension:

This study is optional and will be conducted in patients already enrolled in the "Evaluation and Treatment of Autonomic Failure" and the medication trial part of this protocol. A separate consent form (addendum) will be provided. In the present study, we propose the following:

1. Monitor BP and HR in patients with AF and supine hypertension during a 24-hour period, which includes fixed periods of supine rest during the day, with strict control of physical activities, meals, water ingestion and other confounding factors. This will allow us to learn more about the intrinsic circadian variation of BP in our patients without the influence of "external factors".
2. Characterize the hemodynamic changes underlying the dipping phenomenon and the morning BP surge, and
3. Assess changes in plasma volume (measured by changes in hematocrit), calculated plasma osmolality and hormones that regulate blood pressure and blood volume, in order to learn more about the mechanisms responsible for the dipping phenomenon and morning BP surge in autonomic failure patients with supine hypertension.

These parameters will be compared with the circadian rhythm of body temperature, a marker of the central circadian rhythm, to determine whether these diurnal changes are synchronized to the circadian pacemaker.

The duration of the study day will be 24 hours and can start any time during the day. Typically, the study will start ~ 8AM. Therapeutic trials for orthostatic hypotension and/or supine hypertension as well as other study procedures related to the above mentioned protocols may be performed while participating in this study. If an overnight medication trial is performed during the study, patients may be offered to participate in a second study day without any medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with autonomic failure and with supine hypertension from all races

Exclusion Criteria:

* All medical students
* Pregnant women
* High-risk patients (e.g. heart failure, symptomatic coronary artery disease, liver impairment, history of stroke or myocardial infarction)
* History of serious allergies or asthma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2001-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Decrease in supine systolic blood pressure | 12 hours

SECONDARY OUTCOMES:
Decrease in pressure natriuresis | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Shibao C, Okamoto L, Biaggioni I. Pharmacotherapy of autonomic failure. Pharmacol Ther. 2012 Jun;134(3):279-86. doi: 10.1016/j.pharmthera.2011.05.009. Epub 2011 Jun 12. PMID 21664375
- [Result] Shibao C, Gamboa A, Diedrich A, Biaggioni I. Management of hypertension in the setting of autonomic dysfunction. Curr Treat Options Cardiovasc Med. 2006 Apr;8(2):105-9. doi: 10.1007/s11936-006-0002-1. PMID 16533484
- [Result] Shibao C, Gamboa A, Abraham R, Raj SR, Diedrich A, Black B, Robertson D, Biaggioni I. Clonidine for the treatment of supine hypertension and pressure natriuresis in autonomic failure. Hypertension. 2006 Mar;47(3):522-6. doi: 10.1161/01.HYP.0000199982.71858.11. Epub 2006 Jan 3. PMID 16391172
- [Result] Shibao C, Gamboa A, Diedrich A, Biaggioni I. Management of hypertension in the setting of autonomic failure: a pathophysiological approach. Hypertension. 2005 Apr;45(4):469-76. doi: 10.1161/01.HYP.0000158835.94916.0c. Epub 2005 Feb 28. PMID 15738343
- [Result] Diedrich A, Jordan J, Tank J, Shannon JR, Robertson R, Luft FC, Robertson D, Biaggioni I. The sympathetic nervous system in hypertension: assessment by blood pressure variability and ganglionic blockade. J Hypertens. 2003 Sep;21(9):1677-86. doi: 10.1097/00004872-200309000-00017. PMID 12923400
- [Result] Biaggioni I, Robertson RM. Hypertension in orthostatic hypotension and autonomic dysfunction. Cardiol Clin. 2002 May;20(2):291-301, vii. doi: 10.1016/s0733-8651(01)00005-4. PMID 12119802
- [Result] Jordan J, Biaggioni I. Diagnosis and treatment of supine hypertension in autonomic failure patients with orthostatic hypotension. J Clin Hypertens (Greenwich). 2002 Mar-Apr;4(2):139-45. doi: 10.1111/j.1524-6175.2001.00516.x. PMID 11927799
- [Result] Shannon JR, Jordan J, Diedrich A, Pohar B, Black BK, Robertson D, Biaggioni I. Sympathetically mediated hypertension in autonomic failure. Circulation. 2000 Jun 13;101(23):2710-5. doi: 10.1161/01.cir.101.23.2710. PMID 10851208
- [Result] Jordan J, Shannon JR, Pohar B, Paranjape SY, Robertson D, Robertson RM, Biaggioni I. Contrasting effects of vasodilators on blood pressure and sodium balance in the hypertension of autonomic failure. J Am Soc Nephrol. 1999 Jan;10(1):35-42. doi: 10.1681/ASN.V10135. PMID 9890307
- [Result] Shannon J, Jordan J, Costa F, Robertson RM, Biaggioni I. The hypertension of autonomic failure and its treatment. Hypertension. 1997 Nov;30(5):1062-7. doi: 10.1161/01.hyp.30.5.1062. PMID 9369256
- [Result] Okamoto LE, Gamboa A, Shibao C, Black BK, Diedrich A, Raj SR, Robertson D, Biaggioni I. Nocturnal blood pressure dipping in the hypertension of autonomic failure. Hypertension. 2009 Feb;53(2):363-9. doi: 10.1161/HYPERTENSIONAHA.108.124552. Epub 2008 Dec 1. PMID 19047577
- [Result] Gamboa A, Shibao C, Diedrich A, Paranjape SY, Farley G, Christman B, Raj SR, Robertson D, Biaggioni I. Excessive nitric oxide function and blood pressure regulation in patients with autonomic failure. Hypertension. 2008 Jun;51(6):1531-6. doi: 10.1161/HYPERTENSIONAHA.107.105171. Epub 2008 Apr 21. PMID 18426998
- [Result] Arnold AC, Okamoto LE, Gamboa A, Shibao C, Raj SR, Robertson D, Biaggioni I. Angiotensin II, independent of plasma renin activity, contributes to the hypertension of autonomic failure. Hypertension. 2013 Mar;61(3):701-6. doi: 10.1161/HYPERTENSIONAHA.111.00377. Epub 2012 Dec 24. PMID 23266540
- [Result] Arnold AC, Biaggioni I. Management approaches to hypertension in autonomic failure. Curr Opin Nephrol Hypertens. 2012 Sep;21(5):481-5. doi: 10.1097/MNH.0b013e328356c52f. PMID 22801444
- [Result] Garland EM, Gamboa A, Okamoto L, Raj SR, Black BK, Davis TL, Biaggioni I, Robertson D. Renal impairment of pure autonomic failure. Hypertension. 2009 Nov;54(5):1057-61. doi: 10.1161/HYPERTENSIONAHA.109.136853. Epub 2009 Sep 8. PMID 19738158